CLINICAL TRIAL: NCT00005526
Title: Genetic Basis of Abdominal Aortic Aneurysm
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5058; R01HL044682 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Aortic Aneurysm, Abdominal

SUMMARY:
To identify the genetic (major genes) and environmental factors responsible for the significant aggregation of abdominal aortic aneurysm (AAA) among relatives of affected individuals.

DETAILED DESCRIPTION:
BACKGROUND:

Abdominal aortic aneurysm (AAA) is a dilatation of the abdominal aorta which can, if undetected, lead to rupture. The mortality associated with ruptured AAA is estimated to be 90 percent, while elective repair has a mortality risk of approximately 6 percent. Ruptured AAA is a leading cause of death among older Americans. The identification of markers of AAA risk could lead to preventive intervention. AAA aggregates in families, and segregation analysis shows that familial risk of AAA is best explained by the segregation of a major gene with an autosomal recessive mode of inheritance.

DESIGN NARRATIVE:

Affected relative pairs (primarily sibling pairs) with AAA and no evidence of a family history of a connective tissue disorder were genotyped for 150 highly informative microsatellite polymorphisms marking the autosomal genome at a resolution of 20 cM. The linkage between AAA and these loci was tested using robust affected pedigree member methods to identify genomic regions which might contain genes that predisposed individuals to develop AAA. The existence of predisposing gene(s) were confirmed and their location refined using a defined search strategy, genotyping at increasing levels of resolution, and re-analysis of family data. The predisposing gene(s) were identified by a combination of saturation mapping and molecular analysis of candidate loci. The association of AAA with environmental measures was investigated to determine an equation for estimating risk for relatives of AAA patients based upon environmental measures and genotype. Power calculations based upon the number and structure of families already collected demonstrated the feasibility of identifying genes that predisposed to AAA using this strategy, even in the presence of significant heterogeneity with respect to the loci involved. In addition to identifying genes that were necessary for AAA by linkage analysis, a series of analyses of association were undertaken to identify true susceptibility genes that were neither necessary nor sufficient to cause disease, but which modified an individual's risk of developing AAA.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-08; Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ferrell — University of Pittsburgh

REFERENCES:
- [Background] Peters DG, Kassam A, St Jean PL, Yonas H, Ferrell RE. Functional polymorphism in the matrix metalloproteinase-9 promoter as a potential risk factor for intracranial aneurysm. Stroke. 1999 Dec;30(12):2612-6. doi: 10.1161/01.str.30.12.2612. PMID 10582986
- [Background] Peters DG, Kassam AB, Yonas H, O'Hare EH, Ferrell RE, Brufsky AM. Comprehensive transcript analysis in small quantities of mRNA by SAGE-lite. Nucleic Acids Res. 1999 Dec 15;27(24):e39. doi: 10.1093/nar/27.24.e39. PMID 10572191
- [Background] Vorp DA, Peters DG, Webster MW. Gene expression is altered in perfused arterial segments exposed to cyclic flexure ex vivo. Ann Biomed Eng. 1999 May-Jun;27(3):366-71. doi: 10.1114/1.158. PMID 10374728
- [Background] St Jean P, Hart B, Webster M, Steed D, Adamson J, Powell J, Ferrell R. Alpha-1-antitrypsin deficiency in aneurysmal disease. Hum Hered. 1996 Mar-Apr;46(2):92-7. doi: 10.1159/000154333. PMID 8666418
- [Background] St Jean PL, Zhang XC, Hart BK, Lamlum H, Webster MW, Steed DL, Henney AM, Ferrell RE. Characterization of a dinucleotide repeat in the 92 kDa type IV collagenase gene (CLG4B), localization of CLG4B to chromosome 20 and the role of CLG4B in aortic aneurysmal disease. Ann Hum Genet. 1995 Jan;59(1):17-24. doi: 10.1111/j.1469-1809.1995.tb01602.x. PMID 7762981
- [Background] St Jean PL, Zhang XC, Hart BK, Ferrell RE. Dinucleotide repeat polymorphism at the HPR locus. Hum Mol Genet. 1994 Nov;3(11):2081. No abstract available. PMID 7874138
- [Background] Foster K, Ferrell R, King-Underwood L, Povey S, Attwood J, Rennick R, Humphries SE, Henney AM. Description of a dinucleotide repeat polymorphism in the human elastin gene and its use to confirm assignment of the gene to chromosome 7. Ann Hum Genet. 1993 May;57(2):87-96. doi: 10.1111/j.1469-1809.1993.tb00890.x. PMID 8368807
- [Background] Peters DG, Kassam AB, Feingold E, Heidrich-O'Hare E, Yonas H, Ferrell RE, Brufsky A. Molecular anatomy of an intracranial aneurysm: coordinated expression of genes involved in wound healing and tissue remodeling. Stroke. 2001 Apr;32(4):1036-42. doi: 10.1161/01.str.32.4.1036. PMID 11283408
- [Background] Peters DG, Zhang XC, Benos PV, Heidrich-O'Hare E, Ferrell RE. Genomic analysis of immediate/early response to shear stress in human coronary artery endothelial cells. Physiol Genomics. 2002 Dec 26;12(1):25-33. doi: 10.1152/physiolgenomics.00016.2002. Epub 2002 Dec 26. PMID 12407183